CLINICAL TRIAL: NCT04887311
Title: An Open Label Study to Assess the Safety and Efficacy of MBM-01 for the Treatment of Ataxia Telangiectasia
Brief Title: MBM-01 (Tempol) for the Treatment of Ataxia Telangiectasia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Matrix Biomed, Inc. (Industry)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBI-09-01
Expanded Access: Available
Record Dates: First submitted 2021-05-05; First posted 2021-05-14 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Ataxia Telangiectasia Louis-Bar; Ataxia Telangiectasia in Children; Ataxia Telangiectasia
MeSH Terms: conditions — Ataxia Telangiectasia | interventions — tempol

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Experimental): Group 1 Patients ≥13 years old will receive a total daily dose of 1200 mg/day.
  Group 2 - Group 4
  Patients 4-12 years old will receive group weight-tiered doses at 17 mg/kg:
  Group 2
  * Patients aged 4-12 years weighing 15kg to <25 kg will take 340 mg/day. Group 3
  * Patients aged 4-12 years weighing 25kg to <35 kg will take 510 mg/day. Group 4
  * Patients aged 4-12 years weighing ≥35 kg will take 850 mg/day.
  Interventions: Drug: MBM-01

INTERVENTIONS:
Drug: MBM-01 — Patients will be administered study drug daily for 9 months QD via premarked medicine cups.
  Other Names: Tempol oral solution

SUMMARY:
Ataxia Telangiectasia (A-T) is an autosomal recessively inherited neurodegenerative disorder that also has dramatic effects on the immune and endocrine systems. The disorder results from mutations in the A-T mutated gene (ATM) leading to a loss in the production of the ATM protein.

The active compound in MBM-01 (4-hydroxy-2,2,6,6-tetramethylpiperidine-1-oxyl) may substitute for the loss of ATM by protecting cells from DNA damage, preventing and reducing oxidative damage, triggering an increase in cellular survival proteins, and preserving the brain and peripheral immune system.

DETAILED DESCRIPTION:
Cells lacking ATM are left defenseless and unable to repair cellular damaged DNA, to exhibit normal cell cycle control, to effectively respond to oxidative damage, ionizing radiation, and, alkylating agents, and to maintain a healthy immune response among others. A-T patients have increased oxidative stress and significantly reduced total antioxidant levels. In an early study directed to oxidative stress in A-T patients, a decrease in the levels of total antioxidant capacity has been observed.

There is currently no cure for A-T, and current treatments are limited to palliative care. Therapies include rehabilitative care, infection prevention and treatment, and screening for pulmonary dysfunction and malignancies. Symptomatic treatments generally fall short and leave A-T patients debilitated and in a progressively wasting state. Patients suffering from A-T are in dire need of a treatment to alleviate the conditions of this disease. A drug product that can substitute for the loss of ATM has the potential to provide these patients with this critically unmet need. The active compound in MBM-01 has been shown to supplant the overall role of ATM by reducing oxidative stress, reducing DNA double strand breaks, and decreasing programmed cell death (in healthy cells). Accordingly, MBM-01 represents a potential breakthrough therapy for patients afflicted with A-T providing a multifactorial approached as evidenced by the following:

1. Doubling the lifespan of otherwise short lived ATM-deficient mice ;
2. Increasing NAD+, thereby decreasing the premature aging of A-T patients by reducing the severity of A-T neuropathology, normalizing neuromuscular function, delaying memory loss, and extending lifespan;
3. Increasing the transcription factor BDNF and NRF2 to decrease neurodegeneration and activate cellular defense machinery via antioxidant genes;
4. Maintaining and improving immune system function to ameliorate A-T symptoms ;
5. Protecting DNA from damage and repairing the type of DNA damage observed in A-T patients;
6. Preventing and reducing the type of oxidative stress observed in A-T patients;
7. Increasing the lifespan of mice under various conditions and toxicities; and
8. Decreasing tumorigenesis and carcinogenesis in general.

The study is a multi-center open label study to assess the efficacy of MBM-01 to treat ataxia telangiectasia. Patients will be assessed during three study phases: a baseline period, a 9-month treatment period, and a 3-month follow-up period. Patients will visit sites day 0, month 3, month 6, and month 9 for safety labs and efficacy assessments.

Dosing will follow a weight-tiered dosing schedule administered orally QD via premarked medicine cups. Patients will be administered study drug daily, 7-days a week. The patients will be placed into one of four dosing groups.

ELIGIBILITY:
Inclusion Criteria:

1. Have a confirmed diagnosis of A-T.

   a) Patients will either have a prior molecular confirmation or will be investigated;
2. If female and of childbearing potential, must be using an effective birth-control method with a history of reliability for the individual patient;
3. If a female with a male partner. If the male is of childbearing potential, adequate methods of contraception must be employed including use of condoms with spermicide. No sperm donation for 90 days until after the conclusion of the study;
4. Body weight > 15 kg;
5. Be able to participate for the full term of the clinical investigation;
6. The patient and his/her parent/caregiver (if below the age of consent), or a legal representative, has provided written informed consent to participate. If consent is provided solely by the caregiver in accordance with local regulations, the patient must provide assent to participate in the study

Exclusion Criteria:

1. Females that are

   a) pregnant, or are breast-feeding;
2. Females of childbearing potential who do not use adequate birth control, as determined by their Health Care Provider;
3. Patients with severe vision or hearing impairment (that is not corrected by glasses or hearing aids) that, at the investigator's discretion, interferes with their ability to perform study assessments;
4. Patients who have been diagnosed with arthritis or other musculoskeletal disorders affecting joints, muscles, ligaments, and/or nerves that by themselves affects patient's mobility and, at the investigator's discretion, interferes with their ability to perform study assessments;
5. A disability that may prevent the patient from completing all study requirements;
6. Severe or unstable pulmonary disease;
7. Uncontrolled diabetes. Patients with diabetes that has been stabilized (i.e. no hypoglycemic or hyperglycemic episodes in the past 3 months) will be eligible;
8. Current neoplastic disease or previous neoplastic disease not in remission for at least 2 years;
9. Has participated in any other trial with an investigational drug and received a dose within 30 days;
10. Requires any concomitant medication prohibited by the protocol;
11. Any other severe, unstable, or serious disease or condition that in the Investigator's opinion would put the patient at risk for imminent life-threatening morbidity, need for hospitalization, or mortality; and
12. Evidence of significant medical illness, or psychiatric illness/social situation that would, in the investigator's judgment, make the patient inappropriate for this study.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in International Cooperative Ataxia Rating Scale (ICARS) | ICARS evaluations will be taken at baseline, month 3, month 6, and month 9.
  The ICARS is a 19 item rating scale of ataxia with the total score ranging from 0 to 100. A score of 0 means normal and higher scores represent worsened disease.

SECONDARY OUTCOMES:
Change in Nine Hole Peg Test (9HPT) Baseline (Day 1) to end of treatment with MBM-01 | The change in 9HPT will be taken at baseline, month 3, month 6, and month 9.
Change in Timed 25 Feet Walking Test (T25FW) | T25FW will be assessed at baseline, month 3, month 6, and month 9.
  The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time, in seconds, is calculated from the initiation of the instruction to start and ends when the patient has reached the 25-foot mark. Baseline values are recorded twice.
Change in total antioxidant capacity | (TEAC) taken at baseline, month 3, month 6, and month 9
  The plasma antioxidant capacity will be determined by the trolox-equivalent antioxidant capacity test (TEAC)
Change in Total Plasma Lipid Peroxides | Change in total plasma lipid peroxide levels taken at baseline, month 3, month 6, and month 9.
Change in GSH/glutathione Disulfide (GSSG) Concentration Ratio | taken at baseline, month 3, month 6, and month 9.
  GSH concentrations will be compared to glutathione disulfide.
Change in lymphocyte counts (CD3) | Change in serum lymphocyte counts (CD3) taken at baseline, month 3, month 6, and month 9
Change in lymphocyte counts (CD4) | Change in serum lymphocyte counts (CD4) taken at baseline, month 3, month 6, and month 9
Change in lymphocyte counts (CD8) | Change in serum lymphocyte counts (CD8) taken at baseline, month 3, month 6, and month 9
Change in lymphocyte counts (CD19) | Change in serum lymphocyte counts (CD19) taken at baseline, month 3, month 6, and month 9
Change 8-hydroxy-2- Deoxyguanosine (8-OHdG) | Taken at baseline, month 3, month 6, and month 9.
  Evaluation of 8-hydroxy-2'-deoxyguanosine (8-OHdG) adduct levels in human peripheral blood lymphocytes taken at baseline, month 3, month 6, and month 9.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schubert R, Erker L, Barlow C, Yakushiji H, Larson D, Russo A, Mitchell JB, Wynshaw-Boris A. Cancer chemoprevention by the antioxidant tempol in Atm-deficient mice. Hum Mol Genet. 2004 Aug 15;13(16):1793-802. doi: 10.1093/hmg/ddh189. Epub 2004 Jun 22. PMID 15213104
- See also: Related Info — http://matrixbiomed.com